CLINICAL TRIAL: NCT04058067
Title: A One-Year, Randomized, Double-Masked, Multicenter, Phase III, Two-Arm Study Assessing the Efficacy and Safety of Brolucizumab Versus Aflibercept in Adult Chinese Patients With Visual Impairment Due to Diabetic Macular Edema
Brief Title: To Compare Brolucizumab to Aflibercept in Chinese Patients With Visual Impairment Due to Diabetic Macular Edema
Acronym: KINGLET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRTH258B2304
Record Dates: First submitted 2019-08-14; First posted 2019-08-15 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular edema (DME); Intravitreal injection; brolucizumab; aflibercept; macular edema; diabetic retinopathy
MeSH Terms: conditions — Macular Edema; Diabetic Retinopathy | interventions — brolucizumab; aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brolucizumab 6 mg (Experimental): 5 x every 6 weeks loading then every 12 weeks or every 8 weeks maintenance
  Interventions: Drug: Brolucizumab
- Aflibercept 2 mg (Active Comparator): 5 x every 4 weeks loading then every 8 weeks maintenance
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Brolucizumab — 5 x every 6 weeks loading then every 12 weeks or every 8 weeks maintenance
  Other Names: RTH258
  Arms: Brolucizumab 6 mg
Drug: Aflibercept — 5 x every 4 weeks loading then every 8 weeks maintenance
  Other Names: Eylea
  Arms: Aflibercept 2 mg

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of brolucizumab in treatment of Chinese patients with visual impairment due to Diabetic Macular Edema.

DETAILED DESCRIPTION:
The study is a randomized, double-masked, multi-center, active-controlled, 2-arm study in Chinese patients with Diabetic macular edema (DME). Approximately 335 Chinese patients were planned to be screened (20% screening failure rate expected) and approximately 268 (134 per arm) patients were planned to be randomized in approximately 25 centers.

Patients who met all the inclusion and none of the exclusion criteria were randomized in a 1:1 ratio to one of two treatment arms:

* Brolucizumab 6 mg: 5 × every 6 weeks (q6w) loading then every 12 weeks (q12w) or every 8 weeks (q8w) maintenance
* Aflibercept 2 mg: 5 × every 4 weeks (q4w) loading then q8w maintenance

Disease activity assessments (DAAs) were conducted by the masked investigator for both treatment arms at Weeks 32, 36, and 48. In the brolucizumab arm, subjects who qualified for q12w during this initial q12w interval continued on a q12w treatment frequency unless disease activity was identified at the subsequent DAA visit at Week 48, in which case subjects were switched to a q8w treatment interval until Week 52.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study.
2. Patients ≥18 years of age at screening
3. Patients with type 1 or type 2 diabetes mellitus (DM) and Hemoglobin A1c (HbA1c) of ≤10% at screening
4. Medication for the management of diabetes must have been stable within 3 months prior to randomization and is expected to remain as stable as medically acceptable during the course of the study
5. Study Eye Visual impairment due to diabetic macular edema (DME) with:

   * Best-corrected visual acuity (BCVA) score between 78 and 23 letters, inclusive, using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity (VA) testing charts at a starting testing distance of 4 meters (approximate Snellen equivalent of 20/32 to 20/320) at screening and baseline
   * DME involving the center of the macula, with central subfield retinal thickness (e.g. measured from retinal pigment epithelium (RPE) to the inner limiting membrane (ILM) inclusively) of ≥320 μm on Spectral domain optical coherence tomography (SD-OCT) at screening.

Exclusion Criteria:

* Active Proliferative diabetic retinopathy (PDR) in the study eye as per investigator
* Concomitant conditions or ocular disorders in the study eye at screening or baseline which could, in the opinion of the investigator, prevent response to study treatment or may confound interpretation of study results, compromise visual acuity or require medical or surgical intervention for the duration of the study (e.g. cataract, vitreous hemorrhage, retinal vascular occlusion, retinal detachment, macular hole, or choroidal neovascularization (CNV) of any cause)
* Any active intraocular or periocular infection or active intraocular inflammation (e.g. infectious conjunctivitis, keratitis, scleritis, endophthalmitis, infectious blepharitis, uveitis) in study eye at screening or baseline
* Structural damage of the fovea in the study eye at screening likely to preclude improvement in visual acuity following the resolution of macular edema (ME), including atrophy of the retinal pigment epithelium, subretinal fibrosis, laser scar(s), epiretinal membrane involving fovea or organized hard exudate plaques
* Uncontrolled glaucoma in the study eye defined as intraocular pressure (IOP) > 25 mmHg on medication or according to investigator's judgment at Screening or Baseline
* Neovascularization of the iris in the study eye at screening or baseline
* Evidence of vitreomacular traction in the study eye at screening or baseline which in the opinion of the investigator, affects visual acuity
* Previous treatment with any anti-vascular growth factor (VEGF) drug or investigational drugs in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- China (15):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shantou, Guangdong
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Wuxi, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Qingdao, Shandong
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Nanjing
  - Novartis Investigative Site, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://clinicalstudydatarequest.com/

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1867

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Started | 132 | 131
Completed | 120 | 120
Not Completed | 12 | 11
Not completed — Adverse Event | 2 | 0
Not completed — Death | 0 | 1
Not completed — Physician Decision | 3 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg | Total
Number analyzed (Participants) | 132 | 131 | 263
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 85 | 88 | 173
  >=65 years | 47 | 43 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (9.20) | 58.7 (9.92) | 59.6 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 60 | 122
  Male | 70 | 71 | 141
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 132 | 131 | 263
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 52 in Best-corrected Visual Acuity (BCVA) for the Study Eye.
Description: BCVA was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  Visual Function of the study eye was assessed using the ETDRS protocol.
  Min and max possible scores are 0-100 respectively. A higher score represents better visual functioning.
Time Frame: Baseline to Week 52
Population: Full Analysis Set- last observation carried forward (FAS - LOCF)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
Scores on a scale | 10.6 (0.85) | 11.9 (0.85)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority; p = 0.013, ANOVA; LS mean difference = -1.3, 95% CI 2-sided [-3.7 to 1.1], Standard Error of Mean 1.20

2. Primary Outcome: Best-corrected Visual Acuity (BCVA) - Average Change From Baseline Over the Period Week 40 Through Week 52 for the Study Eye
Description: as for outcome 1
Time Frame: Week 40 to Week 52
Population: Full Analysis Set- last observation carried forward (FAS - LOCF)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
Scores on a scale | 10.1 (0.81) | 12.0 (0.82)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority; p = 0.035, ANOVA; LS mean difference = -1.9, 95% CI 2-sided [-4.2 to 0.4], Standard Error of Mean 1.15

3. Secondary Outcome: Change From Baseline by Visit up to Week 52 in Best-corrected Visual Acuity (BCVA) for the Study Eye
Description: as for outcome 1
Time Frame: Baseline, Week 52
Population: Full Analysis Set- observed. All randomized subjects who received at least one intravitreal treatment (IVT) injection of the study treatment and had a valid value of the outcome measure at each timepoint.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
Scores on a scale
  Week 4 (n=129,123): number analyzed (Participants) | 129 | 123
  Week 4 (n=129,123) | 5.1 (6.58) | 4.4 (6.75)
  Week 6 (n=125,122): number analyzed (Participants) | 125 | 122
  Week 6 (n=125,122) | 7.2 (7.49) | 6.6 (7.50)
  Week 8 (n=128,125): number analyzed (Participants) | 128 | 125
  Week 8 (n=128,125) | 8.6 (8.43) | 8.0 (8.56)
  Week 12 (n=119,122): number analyzed (Participants) | 119 | 122
  Week 12 (n=119,122) | 9.2 (8.77) | 9.0 (9.67)
  Week 16 (n=115,118): number analyzed (Participants) | 115 | 118
  Week 16 (n=115,118) | 10.0 (9.83) | 10.4 (9.86)
  Week 18 (n=113,115): number analyzed (Participants) | 113 | 115
  Week 18 (n=113,115) | 9.8 (9.19) | 10.7 (10.25)
  Week 20 (n=109,114): number analyzed (Participants) | 109 | 114
  Week 20 (n=109,114) | 10.0 (9.36) | 11.3 (9.57)
  Week 24 (n=109,116): number analyzed (Participants) | 109 | 116
  Week 24 (n=109,116) | 9.9 (10.48) | 10.5 (9.80)
  Week 28 (n=111,111): number analyzed (Participants) | 111 | 111
  Week 28 (n=111,111) | 10.5 (9.62) | 10.9 (10.13)
  Week 32 (n=107,116): number analyzed (Participants) | 107 | 116
  Week 32 (n=107,116) | 10.1 (10.29) | 11.3 (10.12)
  Week 36 (n=105,114): number analyzed (Participants) | 105 | 114
  Week 36 (n=105,114) | 9.1 (10.86) | 11.8 (10.62)
  Week 40 (n=101,110): number analyzed (Participants) | 101 | 110
  Week 40 (n=101,110) | 10.1 (10.24) | 11.7 (10.02)
  Week 44 (n=102,110): number analyzed (Participants) | 102 | 110
  Week 44 (n=102,110) | 11.2 (9.86) | 12.2 (9.79)
  Week 48 (n=103,105): number analyzed (Participants) | 103 | 105
  Week 48 (n=103,105) | 10.9 (9.91) | 12.2 (10.71)
  Week 52 (n=105,105): number analyzed (Participants) | 105 | 105
  Week 52 (n=105,105) | 11.3 (9.21) | 12.1 (10.92)

4. Secondary Outcome: Best-corrected Visual Acuity (BCVA) - Average Change From Baseline Over the Period Week 4 Through Week 52 for the Study Eye
Description: as for outcome 1
Time Frame: Week 4 to Week 52
Population: Full Analysis Set- last observation carried forward (FAS - LOCF)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
Scores on a scale | 9.0 (0.68) | 10.1 (0.68)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority; ANOVA; Difference = -1.1, 95% CI 2-sided [-3.0 to 0.8], Standard Error of Mean 0.96

5. Secondary Outcome: Best-corrected Visual Acuity (BCVA) - Average Change From Baseline Over the Period Week 20 Through Week 52 for the Study Eye
Description: as for outcome 1
Time Frame: Week 20 to Week 52
Population: Full Analysis Set- last observation carried forward (FAS - LOCF)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
Scores on a scale | 9.6 (0.77) | 11.5 (0.77)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority; ANOVA; Difference = -1.9, 95% CI 2-sided [-4.0 to 0.2], Standard Error of Mean 1.09

6. Secondary Outcome: Best-corrected Visual Acuity (BCVA) - Average Change From Baseline Over the Period Week 28 Through Week 52 for the Study Eye
Description: as for outcome 1
Time Frame: Week 28 to Week 52
Population: Full Analysis Set- last observation carried forward (FAS - LOCF)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
Scores on a scale | 9.6 (0.80) | 11.7 (0.80)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority; ANOVA; Difference = -2.0, 95% CI 2-sided [-4.3 to 0.2], Standard Error of Mean 1.14

7. Secondary Outcome: Time-to-first q8w Treatment Need: Summary for Brolucizumab Subjects by Disease Activity Assessment Visit
Description: The estimate for the proportion of subjects with a positive q12w treatment status was derived from Kaplan Meier time-to-event analyses for the event 'first q8w-need', applying a 'q8w-need' allocation in case of missing or confounded data attributable to lack of efficacy and/or lack of safety. As a result, the probability that subjects in brolucizumab arm do not need a q8w treatment (and therefore are maintained on a q12w treatment) up to the visit is reported in the table.
Time Frame: Baseline (Week 0), Week 32, Week 36 and Week 48
Population: FAS - Efficacy/Safety approach
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 0
Probability
  Week 0 | 1 [NA to NA] — Not applicable for probability of 1 |
  Week 32 (n=86,0): number analyzed (Participants) | 86 | 0
  Week 32 (n=86,0) | 0.733 [0.626 to 0.813] |
  Week36 (n=59,0): number analyzed (Participants) | 59 | 0
  Week36 (n=59,0) | 0.447 [0.338 to 0.550] |
  Week48 (n=30,0): number analyzed (Participants) | 30 | 0
  Week48 (n=30,0) | 0.417 [0.309 to 0.522] |

8. Secondary Outcome: Time-to-first q8w Treatment Need: Summary for Brolucizumab Subjects by Disease Activity Assessment Visit, Within Those Subjects With no q8w-need During the Initial q12w Cycle
Description: as for outcome 7
Time Frame: Week 36 and Week 48
Population: FAS - Efficacy/Safety approach. Participants in the Full Analysis Set with no identified q8w-need at Week 32 and Week 36.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 35 | 0
Probability
  Week36 (n=35,0) | 1 [NA to NA] — Not applicable for probability of 1 |
  Week48 (n=29,0): number analyzed (Participants) | 29 | 0
  Week48 (n=29,0) | 0.931 [0.751 to 0.982] |

9. Secondary Outcome: Number and Percentage of Patients Who Gained in ≥5, ≥10 and ≥15 ETDRS Letters in BCVA From Baseline to Week 52 for the Study Eye
Description: as for outcome 1
Time Frame: Baseline, Week 52
Population: Full Analysis Set- last observation carried forward (FAS - LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
Participants
  N (%) of subjects with ≥5 letters gain from baseline or reached BCVA of ≥84 letters at Week 52 | 102 | 104
  N (%) of subjects with ≥10 letters gain from baseline or reached BCVA of ≥84 letters at Week 52 | 74 | 76
  N (%) of subjects with ≥15 letters gain from baseline or reached BCVA of ≥84 letters at Week 52 | 44 | 48
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Proportion of subjects with ≥5 letters gain from baseline or reached BCVA of ≥84 letters at Week 52; Test type: Superiority; Regression, Logistic; DIfference = -3.0, 95% CI 2-sided [-13.7 to 6.7]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Proportion of subjects with ≥10 letters gain from baseline or reached BCVA of ≥84 letters at Week 52; Test type: Superiority; Regression, Logistic; Difference = -2.6, 95% CI 2-sided [-14.7 to 9.4]
Statistical Analysis 3: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Proportion of subjects with ≥15 letters gain from baseline or reached BCVA of ≥84 letters at Week 52; Test type: Superiority; Regression, Logistic; Difference = -3.8, 95% CI 2-sided [-15.5 to 6.9]

10. Secondary Outcome: Time to Achieve Gain of >= 5 Letters in BCVA From Baseline or Reach BCVA >=84 Letters for the Study Eye - Probability of BCVA Gain
Description: as for outcome 1
Time Frame: Baseline up to Week 52
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Probability of BCVA gain
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
Probability of BCVA gain
  Week 4 | 0.136 [0.084 to 0.201] | 0.038 [0.014 to 0.081]
  Week 6 (n=114,126): number analyzed (Participants) | 114 | 126
  Week 6 (n=114,126) | 0.508 [0.419 to 0.589] | 0.420 [0.334 to 0.503]
  Week 8 (n=65, 76): number analyzed (Participants) | 65 | 76
  Week 8 (n=65, 76) | 0.720 [0.634 to 0.789] | 0.634 [0.544 to 0.710]
  Week 12 (n=37, 48): number analyzed (Participants) | 37 | 48
  Week 12 (n=37, 48) | 0.780 [0.699 to 0.842] | 0.725 [0.639 to 0.794]
  Week 16 (n=29, 36): number analyzed (Participants) | 29 | 36
  Week 16 (n=29, 36) | 0.818 [0.740 to 0.875] | 0.780 [0.697 to 0.842]
  Week 18 (n=24, 28): number analyzed (Participants) | 24 | 28
  Week 18 (n=24, 28) | 0.818 [0.740 to 0.875] | 0.843 [0.766 to 0.896]
  Week 20 (n=24,20): number analyzed (Participants) | 24 | 20
  Week 20 (n=24,20) | 0.841 [0.765 to 0.894] | 0.866 [0.793 to 0.915]
  Week 24 (n=21,17): number analyzed (Participants) | 21 | 17
  Week 24 (n=21,17) | 0.856 [0.782 to 0.906] | 0.874 [0.802 to 0.921]
  Week 28 (n=19,15): number analyzed (Participants) | 19 | 15
  Week 28 (n=19,15) | 0.864 [0.791 to 0.913] | 0.882 [0.811 to 0.928]
  Week 32 (n=17,14): number analyzed (Participants) | 17 | 14
  Week 32 (n=17,14) | 0.888 [0.818 to 0.932] | 0.882 [0.811 to 0.928]
  Week 36 (n=14,14,): number analyzed (Participants) | 14 | 14
  Week 36 (n=14,14,) | 0.888 [0.818 to 0.932] | 0.882 [0.811 to 0.928]
  Week 40 (n=14,14): number analyzed (Participants) | 14 | 14
  Week 40 (n=14,14) | 0.888 [0.818 to 0.932] | 0.908 [0.840 to 0.948]
  Week 44 (n=14,11): number analyzed (Participants) | 14 | 11
  Week 44 (n=14,11) | 0.896 [0.828 to 0.938] | 0.908 [0.840 to 0.948]
  Week 48 (n=13,10): number analyzed (Participants) | 13 | 10
  Week 48 (n=13,10) | 0.912 [0.846 to 0.951] | 0.917 [0.850 to 0.955]
  Week 52 (n=11,9): number analyzed (Participants) | 11 | 9
  Week 52 (n=11,9) | 0.957 [0.880 to 0.985] | 0.926 [0.860 to 0.962]

11. Secondary Outcome: Time to Achieve Gain of >= 10 Letters in BCVA From Baseline or Reach BCVA >=84 Letters for the Study Eye - Probability of BCVA Gain
Description: as for outcome 1
Time Frame: Baseline up to Week 52
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Probability of BCVA gain
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
Probability of BCVA gain
  Week 4 | 0.061 [0.028 to 0.110] | 0.000 [NA to NA] — CI is NA when probability is 0.
  Week 6 (n=124,131): number analyzed (Participants) | 124 | 131
  Week 6 (n=124,131) | 0.227 [0.160 to 0.302] | 0.198 [0.135 to 0.271]
  Week 8 (n=102,105): number analyzed (Participants) | 102 | 105
  Week 8 (n=102,105) | 0.394 [0.310 to 0.476] | 0.306 [0.229 to 0.386]
  Week 12 (n=80,90): number analyzed (Participants) | 80 | 90
  Week 12 (n=80,90) | 0.508 [0.419 to 0.590] | 0.439 [0.352 to 0.523]
  Week 16 (n=64,71): number analyzed (Participants) | 64 | 71
  Week 16 (n=64,71) | 0.562 [0.472 to 0.642] | 0.527 [0.436 to 0.609]
  Week 18 (n=55,59): number analyzed (Participants) | 55 | 59
  Week 18 (n=55,59) | 0.594 [0.504 to 0.673] | 0.551 [0.460 to 0.633]
  Week 20 (n=50,56): number analyzed (Participants) | 50 | 56
  Week 20 (n=50,56) | 0.618 [0.528 to 0.696] | 0.591 [0.500 to 0.671]
  Week 24 (n=47,51): number analyzed (Participants) | 47 | 51
  Week 24 (n=47,51) | 0.643 [0.553 to 0.719] | 0.664 [0.573 to 0.739]
  Week 28 (n=44,41): number analyzed (Participants) | 44 | 41
  Week 28 (n=44,41) | 0.659 [0.570 to 0.735] | 0.680 [0.590 to 0.754]
  Week 32 (n=41,38): number analyzed (Participants) | 41 | 38
  Week 32 (n=41,38) | 0.676 [0.587 to 0.750] | 0.705 [0.616 to 0.777]
  Week 36 (n=39,35): number analyzed (Participants) | 39 | 35
  Week 36 (n=39,35) | 0.693 [0.604 to 0.766] | 0.722 [0.634 to 0.793]
  Week 40 (n=35,33): number analyzed (Participants) | 35 | 33
  Week 40 (n=35,33) | 0.710 [0.622 to 0.782] | 0.730 [0.642 to 0.800]
  Week 44 (n=33,32): number analyzed (Participants) | 33 | 32
  Week 44 (n=33,32) | 0.728 [0.640 to 0.798] | 0.739 [0.652 to 0.808]
  Week 48 (n=31,28): number analyzed (Participants) | 31 | 28
  Week 48 (n=31,28) | 0.754 [0.667 to 0.822] | 0.749 [0.661 to 0.817]
  Week 52 (n=28,27): number analyzed (Participants) | 28 | 27
  Week 52 (n=28,27) | 0.899 [0.416 to 0.987] | 1 [NA to NA] — CI is NA when probability = 1.

12. Secondary Outcome: Time to Achieve Gain of >= 15 Letters in BCVA From Baseline or Reach BCVA >=84 Letters for the Study Eye - Probability of BCVA Gain
Description: as for outcome 1
Time Frame: Baseline up to Week 52
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Probability of BCVA gain
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
Probability of BCVA gain
  Week 4 | 0.008 [0.001 to 0.038] | 0.000 [NA to NA] — CI is NA when probability = 0.
  Week 6 (n=131,131): number analyzed (Participants) | 131 | 131
  Week 6 (n=131,131) | 0.083 [0.044 to 0.138] | 0.069 [0.034 to 0.121]
  Week 8 (n=121,122): number analyzed (Participants) | 121 | 122
  Week 8 (n=121,122) | 0.152 [0.096 to 0.218] | 0.161 [0.104 to 0.229]
  Week 12 (n=112,109): number analyzed (Participants) | 112 | 109
  Week 12 (n=112,109) | 0.227 [0.160 to 0.302] | 0.216 [0.149 to 0.290]
  Week 16 (n=101,100): number analyzed (Participants) | 101 | 100
  Week 16 (n=101,100) | 0.266 [0.193 to 0.343] | 0.255 [0.183 to 0.333]
  Week 18 (n=94,94): number analyzed (Participants) | 94 | 94
  Week 18 (n=94,94) | 0.313 [0.235 to 0.393] | 0.319 [0.240 to 0.401]
  Week 20 (n=87,85): number analyzed (Participants) | 87 | 85
  Week 20 (n=87,85) | 0.344 [0.264 to 0.426] | 0.359 [0.276 to 0.442]
  Week 24 (n=82,80): number analyzed (Participants) | 82 | 80
  Week 24 (n=82,80) | 0.409 [0.323 to 0.492] | 0.399 [0.313 to 0.483]
  Week 28 (n=72,74): number analyzed (Participants) | 72 | 74
  Week 28 (n=72,74) | 0.425 [0.338 to 0.509] | 0.432 [0.344 to 0.516]
  Week 32 (n=67,69): number analyzed (Participants) | 67 | 69
  Week 32 (n=67,69) | 0.459 [0.370 to 0.544] | 0.456 [0.367 to 0.541]
  Week 36 (n=63,66): number analyzed (Participants) | 63 | 66
  Week 36 (n=63,66) | 0.485 [0.395 to 0.570] | 0.481 [0.391 to 0.566]
  Week 40 (n=58,63): number analyzed (Participants) | 58 | 63
  Week 40 (n=58,63) | 0.494 [0.403 to 0.579] | 0.506 [0.415 to 0.590]
  Week 44 (n=57,60): number analyzed (Participants) | 57 | 60
  Week 44 (n=57,60) | 0.512 [0.420 to 0.596] | 0.531 [0.439 to 0.614]
  Week 48 (n=55,54): number analyzed (Participants) | 55 | 54
  Week 48 (n=55,54) | 0.539 [0.446 to 0.622] | 0.540 [0.447 to 0.623]
  Week 52 (n=52,53): number analyzed (Participants) | 52 | 53
  Week 52 (n=52,53) | 0.623 [0.436 to 0.763] | 1 [NA to NA] — CI is NA when probability = 1.

13. Secondary Outcome: Number and Percentage of Patients Who Lost ≥5, ≥10 and ≥15 ETDRS Letters in BCVA From Baseline to Week 52 for the Study Eye
Description: as for outcome 1
Time Frame: Baseline, Week 52
Population: Full Analysis Set- last observation carried forward (FAS - LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
Participants
  N (%) of subjects with ≥5 letters loss from baseline or reached BCVA of ≥84 letters at Week 52 | 4 | 4
  N (%) of subjects with ≥10 letters loss from baseline or reached BCVA of ≥84 letters at Week 52 | 2 | 1
  N (%) of subjects with ≥15 letters loss from baseline or reached BCVA of ≥84 letters at Week 52 | 1 | 1
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Proportion of subjects with ≥5 letters loss from baseline at Week 52; Test type: Superiority; Regression, Logistic; DIfference = 0.1, 95% CI 2-sided [-4.2 to 4.4]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Proportion of subjects with ≥10 letters loss from baseline at Week 52; Test type: Superiority; Regression, Logistic; Difference = 0.8, 95% CI 2-sided [-1.6 to 3.8]
Statistical Analysis 3: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Proportion of subjects with ≥15 letters loss from baseline at Week 52; Test type: Superiority; Regression, Logistic; Difference = 0.0, 95% CI 2-sided [-2.2 to 2.3]

14. Secondary Outcome: Proportion of Patients Who Have Absolute BCVA ≥73 ETDRS Letters at Each Post-baseline Visit for the Study Eye
Description: as for outcome 1
Time Frame: Baseline up to Week 52
Population: Full Analysis Set - LOCF
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
Participants
  Week 4 | 32 | 34
  Week 6 | 36 | 46
  Week 8 | 46 | 55
  Week 12 | 50 | 63
  Week 16 | 50 | 67
  Week 18 | 51 | 68
  Week 20 | 54 | 65
  Week 24 | 53 | 74
  Week 28 | 52 | 72
  Week 32 | 51 | 74
  Week 36 | 49 | 77
  Week 40 | 53 | 81
  Week 44 | 53 | 76
  Week 48 | 57 | 78
  Week 52 | 55 | 75
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 4; Test type: Other — Descriptive, Week 4; Clopper-Pearson exact method; Difference - % = 0.4, 95% CI 2-sided [-7.9 to 8.6]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 6; Test type: Other — Descriptive, Week 6; Clopper-Pearson exact method; Difference - % = -5.1, 95% CI 2-sided [-14.3 to 2.9]
Statistical Analysis 3: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 8; Test type: Other — Descriptive, Week 8; Clopper-Pearson exact method; Difference - % = -4.0, 95% CI [-13.3 to 4.4]
Statistical Analysis 4: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 12; Test type: Other — Descriptive, Week 12; Clopper-Pearson exact method; Difference - % = -7.0, 95% CI 2-sided [-16.4 to 2.3]
Statistical Analysis 5: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 16; Test type: Other — Descriptive, Week 16; Clopper-Pearson exact method; Difference - % = -9.8, 95% CI 2-sided [-19.2 to -0.0]
Statistical Analysis 6: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 18; Test type: Other — Descriptive, Week 18; Clopper-Pearson exact method; Difference - % = -9.8, 95% CI 2-sided [-19.0 to -0.0]
Statistical Analysis 7: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 20; Test type: Other — Descriptive, Week 20; Clopper-Pearson exact method; Difference - % = -5.7, 95% CI 2-sided [-15.8 to 3.9]
Statistical Analysis 8: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 24; Test type: Other — Descriptive, Week 24; Clopper-Pearson exact method; Difference - % = -13.4, 95% CI 2-sided [-23.9 to -3.1]
Statistical Analysis 9: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 28; Test type: Other — Descriptive, Week 28; Clopper-Pearson exact method; Difference - % = -12.4, 95% CI 2-sided [-22.0 to -2.1]
Statistical Analysis 10: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 32; Test type: Other — Descriptive, Week 32; Clopper-Pearson exact method; Difference - % = -15.4, 95% CI 2-sided [-26.0 to -4.8]
Statistical Analysis 11: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 36; Test type: Other — Descriptive, Week 36; Clopper-Pearson exact method; Difference - % = -18.8, 95% CI 2-sided [-29.5 to -8.9]
Statistical Analysis 12: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 40; Test type: Other — Descriptive, Week 40; Clopper-Pearson exact method; Difference - % = -18.4, 95% CI 2-sided [-28.7 to -8.6]
Statistical Analysis 13: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 44; Test type: Other — Descriptive, Week 44; Clopper-Pearson exact method; Difference - % = -14.9, 95% CI 2-sided [-25.6 to -4.4]
Statistical Analysis 14: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 48; Test type: Other — Descriptive, Week 48; Clopper-Pearson exact method; Difference - % = -13.3, 95% CI 2-sided [-23.6 to -3.4]
Statistical Analysis 15: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 52; Test type: Other — Descriptive, Week 52; Clopper-Pearson exact method; Difference - % = -12.6, 95% CI 2-sided [-23.5 to -2.9]

15. Secondary Outcome: Number (%) of Subjects With q8w Treatment Need as Assessed by the Investigator at First Disease Activity Assessment (DAA) Visit - Week 32
Description: To evaluate the efficacy related to dosing regimen of brolucizumab
Time Frame: Week 32
Population: Full Analysis Set - Observed (Patients with a valid observed value for the outcome measure.)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 107 | 115
Participants | 34 | 38
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority; Clopper-Pearson exact method; Difference = -1.3, 95% CI 2-sided [-13.6 to 11.2]

16. Secondary Outcome: Number (%) of Subjects With q8w Treatment Need as Assessed by the Investigator at Week 36, and Week 48
Description: To evaluate the efficacy related to dosing regimen of brolucizumab
Time Frame: Week 36, Week 48
Population: Full Analysis Set - Observed
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 105 | 113
Participants
  Week 36 (n=105,113) | 50 | 32
  Week 48 (n=102,104): number analyzed (Participants) | 102 | 104
  Week 48 (n=102,104) | 25 | 32

17. Secondary Outcome: Change From Baseline at Week 52 in Central Subfield Thickness (CSFT) for the Study Eye
Description: Central Subfield Thickness Assessed by Spectral domain optical coherence tomography (SD-OCT) from the central reading center.
Time Frame: Baseline, Week 52
Population: Full Analysis Set- last observation carried forward (FAS - LOCF)
Measure: Least Squares Mean (Standard Error); unit: micrometer
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
micrometer | -225.2 (9.71) | -215.0 (9.75)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority; ANOVA; Difference = -10.2, 95% CI 2-sided [-37.3 to 17.0], Standard Error of Mean 13.79

18. Secondary Outcome: Average Change From Baseline Over the Period Week 40 Through Week 52 in Central Subfield Thickness (CSFT) for the Study Eye
Description: as for outcome 17
Time Frame: Baseline, over the period of Week 40 to Week 52
Population: Full Analysis Set- last observation carried forward (FAS - LOCF)
Measure: Least Squares Mean (Standard Error); unit: micrometer
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
micrometer | -215.1 (8.69) | -212.7 (8.73)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority; ANOVA; Difference = -2.5, 95% CI 2-sided [-26.8 to 21.9], Standard Error of Mean 12.34

19. Secondary Outcome: Average Change From Baseline Over the Period Week 4 Through Week 52 in Central Subfield Thickness (CSFT) for the Study Eye
Description: as for outcome 17
Time Frame: Baseline, over the period of Week 4 to Week 52
Population: Full Analysis Set- last observation carried forward (FAS - LOCF)
Measure: Least Squares Mean (Standard Error); unit: micrometer
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
micrometer | -207.7 (7.77) | -199.2 (7.80)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority; ANOVA; Difference = -8.5, 95% CI 2-sided [-30.3 to 13.2], Standard Error of Mean 11.03

20. Secondary Outcome: Number and Percentage of Patients Who Have CSFT (<280 Microns) at Each Assessment Visit for the Study Eye
Description: as for outcome 17
Time Frame: Baseline up to Week 52
Population: Full Analysis Set - LOCF
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
Participants
  Week 4 | 24 | 17
  Week 6 | 36 | 22
  Week 8 | 48 | 29
  Week 12 | 52 | 33
  Week 16 | 63 | 41
  Week 18 | 61 | 41
  Week 20 | 67 | 46
  Week 24 | 65 | 40
  Week 28 | 71 | 49
  Week 32 | 63 | 47
  Week 36 | 59 | 51
  Week 40 | 67 | 47
  Week 44 | 74 | 56
  Week 48 | 68 | 52
  Week 52 | 79 | 56
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 4; Test type: Superiority; Clopper-Pearson exact method; Difference - % = 5.3, 95% CI 2-sided [-3.3 to 13.5]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 6; Test type: Superiority; Clopper-Pearson exact method; Difference - % = 10.8, 95% CI 2-sided [1.4 to 20.6]
Statistical Analysis 3: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 8; Test type: Superiority; Clopper-Pearson exact method; Difference - % = 14.1, 95% CI 2-sided [3.9 to 25.3]
Statistical Analysis 4: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 12; Test type: Superiority; Clopper-Pearson exact method; Difference - % = 14.1, 95% CI 2-sided [2.8 to 24.9] — Proportion estimates (%) = 39.3
Statistical Analysis 5: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 16; Test type: Superiority; Clopper-Pearson exact method; Difference - % = 16.8, 95% CI [5.1 to 28.6]
Statistical Analysis 6: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 18; Test type: Superiority; Clopper-Pearson exact method; Difference - % = 15.4, 95% CI 2-sided [3.1 to 26.6]
Statistical Analysis 7: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 20; Test type: Superiority; Clopper-Pearson exact method; Difference - % = 15.7, 95% CI 2-sided [3.5 to 27.1]
Statistical Analysis 8: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 24; Test type: Superiority; Clopper-Pearson exact method; Difference - % = 19.1, 95% CI 2-sided [7.2 to 30.2]
Statistical Analysis 9: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 28; Test type: Superiority; Clopper-Pearson exact method; Difference - % = 16.4, 95% CI 2-sided [4.9 to 27.9]
Statistical Analysis 10: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 32; Test type: Superiority; Clopper-Pearson exact method; Difference - % = 12.1, 95% CI 2-sided [0.4 to 24.4]
Statistical Analysis 11: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 36; Test type: Superiority; Clopper-Pearson exact method; Difference - % = 6.0, 95% CI 2-sided [-5.9 to 18.0]
Statistical Analysis 12: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 40; Test type: Superiority; Clopper-Pearson exact method; Difference - % = 15.2, 95% CI 2-sided [3.3 to 26.1]
Statistical Analysis 13: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 44; Test type: Superiority; Clopper-Pearson exact method; Difference - % = 13.2, 95% CI 2-sided [1.9 to 25.7]
Statistical Analysis 14: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 48; Test type: Superiority; Clopper-Pearson exact method; Difference - % = 11.9, 95% CI 2-sided [-0.8 to 23.6]
Statistical Analysis 15: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 52; Test type: Superiority; Clopper-Pearson exact method; Difference - % = 17.9, 95% CI 2-sided [5.8 to 30.5]

21. Secondary Outcome: Number (%) of Patients With Progression to Proliferative Diabetic Retinopathy (PDR) as Assessed by ETDRS DRSS of at Least 61 by Week 52 for the Study Eye Among the Subset of Non-PDR Subjects at Screening
Description: As evaluated using the Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) score assessed by the Central Reading Center (CRC) based on color fundus photography images in the study eye.
  When the ETDRS-DR severities were evaluable, they were converted and categorized on a 12-level scale, from 1 (DR absent) to 12 (very advanced PDR). A lower score represents better visual functioning.
Time Frame: Baseline, Week 52
Population: Full Analysis Set - LOCF. Subset of non-Proliferative diabetic retinopathy (PDR) subjects at screening
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 106 | 107
Participants | 1 | 0
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority; Clopper-Pearson exact method; Difference = 0.9, 95% CI 2-sided [0.8 to 3.6]

22. Secondary Outcome: Number (%) of Patients With Presence of Leakage in the Study Eye on Fluorescein Angiography (FA)
Description: Assessed by angiography.
Time Frame: Week 52
Population: Full Analysis Set - LOCF
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
Participants | 110 | 115
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority; Clopper-Pearson exact method; Difference = -4.3, 95% CI 2-sided [-13.2 to 4.6]

23. Secondary Outcome: Number (%) of Patients With Presence of Subretinal Fluid (SRF), Intraretinal Fluid (IRF) in the Study Eye
Description: To evaluate the efficacy of brolucizumab relative to aflibercept over the time period by assessing changes in anatomical parameters
Time Frame: Baseline up to Week 52
Population: Full Analysis Set- last observation carried forward (FAS - LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
Participants | 87 | 85
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Superiority; Clopper-Pearson exact method; Difference = 1.0, 95% CI 2-sided [-10.5 to 12.4]

24. Secondary Outcome: Number of Patients With Presence of Subretinal Fluid (SRF) in the Study at Each Assessment Visit
Description: Subretinal Fluid (SRF) status in the central subfield: proportion of subjects with presence of SRF in the study eye by visit
Time Frame: Week 4, 6, 8, 12, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: Full Analysis Set - LOCF
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
Participants
  Week 4 | 33 | 37
  Week 6 | 17 | 28
  Week 8 | 13 | 20
  Week 12 | 7 | 14
  Week 16 | 6 | 9
  Week 18 | 6 | 4
  Week 20 | 6 | 2
  Week 24 | 5 | 2
  Week 28 | 5 | 5
  Week 32 | 8 | 7
  Week 36 | 13 | 8
  Week 40 | 7 | 6
  Week 44 | 7 | 3
  Week 48 | 10 | 4
  Week 52 | 9 | 4

25. Secondary Outcome: Number of Patients With Presence of Intraretinal Fluid (IRF) in the Study at Each Assessment Visit
Description: Intraretinal Fluid (IRF) status in the central subfield: proportion of subjects with presence of IRF in the study eye by visit
Time Frame: Week 4, 6, 8, 12, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: Full Analysis Set - LOCF
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
Participants
  Week 4 | 113 | 115
  Week 6 | 112 | 110
  Week 8 | 109 | 112
  Week 12 | 100 | 110
  Week 16 | 99 | 109
  Week 18 | 98 | 110
  Week 20 | 94 | 102
  Week 24 | 90 | 102
  Week 28 | 87 | 100
  Week 32 | 88 | 99
  Week 36 | 98 | 98
  Week 40 | 89 | 101
  Week 44 | 84 | 94
  Week 48 | 89 | 94
  Week 52 | 87 | 85

26. Secondary Outcome: Intraretinal Fluid (IRF) Status in the Central Subfield: Proportion of Subjects With Presence of IRF in the Study Eye by Visit
Description: Subretinal Fluid (SRF) and Intraretinal Fluid (IRF) status in the central subfield: proportion of subjects with presence of SRF and/or IRF in the study eye by visit
Time Frame: Week 4, 6, 8, 12, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: Full Analysis Set - LOCF
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
Participants
  Week 4 | 117 | 118
  Week 6 | 113 | 114
  Week 8 | 111 | 114
  Week 12 | 100 | 110
  Week 16 | 99 | 110
  Week 18 | 98 | 110
  Week 20 | 94 | 102
  Week 24 | 90 | 102
  Week 28 | 87 | 100
  Week 32 | 88 | 99
  Week 36 | 98 | 98
  Week 40 | 89 | 101
  Week 44 | 84 | 94
  Week 48 | 89 | 94
  Week 52 | 87 | 85

27. Secondary Outcome: Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS): Number of Subjects With >=2-step Improvement From Baseline in the DRSS Score at Each Assessment Visit for the Study Eye - Number of Subjects
Description: Severity of Diabetic Retinopathy (DR) was evaluated using the ETDRS DRSS score assessed by the Central Reading Center (CRC) based on color fundus photography images in the study eye. When the ETDRS-DR severities were evaluable, they were categorized on a 12-level scale, from 1 (DR absent) to 12 (very advanced PDR). A lower score represents better visual functioning.
Time Frame: Baseline, Week 28 and Week 52
Population: FAS - LOCF. For subjects with an assessment of the criterion.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 130
Participants
  Week 28 | 45 | 47
  Week 52 | 62 | 64

28. Secondary Outcome: Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS): Proportion of Subjects With >=2-step Improvement From Baseline in the DRSS Score at Each Assessment Visit for the Study Eye - Percentage Estimates
Description: as for outcome 27
Time Frame: Baseline, Week 28 and Week 52
Population: FAS - LOCF. For subjects with an assessment of the criterion.
Measure: Number; unit: Percentage estimates
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 130
Percentage estimates
  Week 28 | 33.9 | 36.3
  Week 52 | 46.7 | 49.5
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 28; Test type: Other — Descriptive, Week 28; Clopper-Pearson exact method; Difference - % = -2.4, 95% CI 2-sided [-13.9 to 8.8]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 52; Test type: Other — Descriptive, Week 52; Clopper-Pearson exact method; Difference - % = -2.8, 95% CI 2-sided [-14.1 to 9.0]

29. Secondary Outcome: Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS): Number of Subjects With >=3-step Improvement From Baseline in the DRSS Score at Each Assessment Visit for the Study Eye - Number of Subjects
Description: as for outcome 27
Time Frame: Baseline, Week 28 and Week 52
Population: FAS - LOCF. For subjects with an assessment of the criterion.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 130
Participants
  Week 28 | 21 | 15
  Week 52 | 25 | 25

30. Secondary Outcome: Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS): Proportion of Subjects With >=3-step Improvement From Baseline in the DRSS Score at Each Assessment Visit for the Study Eye - Percentage Estimates
Description: as for outcome 27
Time Frame: Baseline, Week 28 and Week 52
Population: FAS - LOCF. For subjects with an assessment of the criterion.
Measure: Number; unit: Percentage estimates
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 130
Percentage estimates
  Week 28 | 15.8 | 11.6
  Week 52 | 18.8 | 19.3
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 28; Test type: Other — Descriptive, Week 28; Clopper-Pearson exact method; Difference - % = 4.2, 95% CI 2-sided [-4.1 to 12.6]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 52; Test type: Other — Descriptive, Week 52; Clopper-Pearson exact method; Difference - % = -0.5, 95% CI 2-sided [-10.5 to 9.3]

31. Secondary Outcome: Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS): Number of Subjects With >=2-step Worsening From Baseline in the DRSS Score at Each Assessment Visit for the Study Eye - Number of Subjects
Description: as for outcome 27
Time Frame: Baseline, Week 28 and Week 52
Population: FAS - LOCF. For subjects with an assessment of the criterion.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 130
Participants
  Week 28 | 1 | 0
  Week 52 | 0 | 0

32. Secondary Outcome: Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS): Proportion of Subjects With >=2-step Worsening From Baseline in the DRSS Score at Each Assessment Visit for the Study Eye - Percentage Estimates
Description: as for outcome 27
Time Frame: Baseline, Week 28 and Week 52
Population: FAS - LOCF. For subjects with an assessment of the criterion.
Measure: Number; unit: Percentage estimates
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 130
Percentage estimates
  Week 28 | 0.8 | 0.0
  Week 52 (n=0,0): number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 28; Test type: Other — Descriptive, Week 28; Clopper-Pearson exact method; Difference - % = 0.8, 95% CI 2-sided [0.7 to 2.9]

33. Secondary Outcome: Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS): Number of Subjects With >=3-step Worsening From Baseline in the DRSS Score at Each Assessment Visit for the Study Eye - Number of Subjects
Description: as for outcome 27
Time Frame: Baseline, Week 28 and Week 52
Population: FAS - LOCF. For subjects with an assessment of the criterion.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 130
Participants
  Week 28 | 1 | 0
  Week 52 | 0 | 0

34. Secondary Outcome: Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS): Proportion of Subjects With >=3-step Worsening From Baseline in the DRSS Score at Each Assessment Visit for the Study Eye - Percentage Estimates
Description: as for outcome 27
Time Frame: Baseline, Week 28 and Week 52
Population: FAS - LOCF. For subjects with an assessment of the criterion.
Measure: Number; unit: Percentage estimates
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 130
Percentage estimates
  Week 28 | 0.8 | 0.0
  Week 52 (n=0,0): number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 28; Test type: Other — Descriptive, Week 28; Clopper-Pearson exact method; Difference - % = 0.8, 95% CI 2-sided [0.7 to 2.9]

35. Secondary Outcome: Change From Baseline at Week 28 and Week 52 in Patient Reported Outcomes (Visual Function Questionnaire-25) - Overall Score
Description: The National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) measures the influence of visual disability and visual symptoms on general health domains.
  The NEI VFQ-25 consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. All items are scored so that a high score represents better visual functioning. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points, respectively. A composite score is derived based on the average of the 11 subscales.
Time Frame: Baseline, Week 28 and Week 52
Population: Full Analysis Set - Observed
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 101 | 103
Scores on a Scale
  Week 28 | 5.3 (11.97) | 7.7 (15.98)
  Week 52 (n=101,101): number analyzed (Participants) | 101 | 101
  Week 52 (n=101,101) | 5.4 (13.87) | 6.6 (16.50)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 28; Test type: Superiority; ANCOVA; LS mean difference = -0.9, 95% CI [-4.1 to 2.3]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 52; Test type: Superiority; ANCOVA; LS mean difference = 0.1, 95% CI 2-sided [-3.1 to 3.3]

36. Secondary Outcome: Change From Baseline at Week 28 and Week 52 in Patient Reported Outcomes (Visual Function Questionnaire-25) - General Vision
Description: as for outcome 35
Time Frame: Baseline, Week 28 and Week 52
Population: Full Analysis Set - Observed
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 101 | 103
Scores on a Scale
  Week 28 (n=96,103): number analyzed (Participants) | 96 | 103
  Week 28 (n=96,103) | 10.4 (18.80) | 9.5 (18.75)
  Week 52 (n=101,101): number analyzed (Participants) | 101 | 101
  Week 52 (n=101,101) | 10.9 (18.23) | 11.5 (17.74)

37. Secondary Outcome: Change From Baseline at Week 28 and Week 52 in Patient Reported Outcomes (Visual Function Questionnaire-25) - Ocular Pain
Description: as for outcome 35
Time Frame: Baseline, Week 28 and Week 52
Population: Full Analysis Set - Observed
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 101 | 103
Scores on a Scale
  Week 28 (n=96,103): number analyzed (Participants) | 96 | 103
  Week 28 (n=96,103) | 5.1 (20.16) | 5.3 (24.23)
  Week 52 (n=101,101): number analyzed (Participants) | 101 | 101
  Week 52 (n=101,101) | 3.5 (22.51) | 2.6 (25.27)

38. Secondary Outcome: Change From Baseline at Week 28 and Week 52 in Patient Reported Outcomes (Visual Function Questionnaire-25) - Near Activities
Description: as for outcome 35
Time Frame: Baseline, Week 28 and Week 52
Population: Full Analysis Set - Observed
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 100 | 103
Scores on a Scale
  Week 28 (n=96,103): number analyzed (Participants) | 96 | 103
  Week 28 (n=96,103) | 8.5 (20.79) | 9.7 (24.15)
  Week 52 (n=100,101): number analyzed (Participants) | 100 | 101
  Week 52 (n=100,101) | 7.8 (22.12) | 8.0 (25.25)

39. Secondary Outcome: Change From Baseline at Week 28 and Week 52 in Patient Reported Outcomes (Visual Function Questionnaire-25) - Distance Activities
Description: as for outcome 35
Time Frame: Baseline, Week 28 and Week 52
Population: Full Analysis Set - Observed
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 101 | 103
Scores on a Scale
  Week 28 (n=96,103): number analyzed (Participants) | 96 | 103
  Week 28 (n=96,103) | 5.6 (17.54) | 7.6 (22.34)
  Week 52 (n=101,101): number analyzed (Participants) | 101 | 101
  Week 52 (n=101,101) | 4.2 (18.42) | 6.5 (22.43)

40. Secondary Outcome: Change From Baseline at Week 28 and Week 52 in Patient Reported Outcomes (Visual Function Questionnaire-25) - Social Functioning
Description: as for outcome 35
Time Frame: Baseline, Week 28 and Week 52
Population: Full Analysis Set - Observed
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 101 | 103
Scores on a Scale
  Week 28 (n=96,103): number analyzed (Participants) | 96 | 103
  Week 28 (n=96,103) | 3.8 (14.86) | 5.2 (18.98)
  Week 52 (n=101,101): number analyzed (Participants) | 101 | 101
  Week 52 (n=101,101) | 3.7 (15.47) | 5.8 (17.73)

41. Secondary Outcome: Change From Baseline at Week 28 and Week 52 in Patient Reported Outcomes (Visual Function Questionnaire-25) - Mental Health
Description: as for outcome 35
Time Frame: Baseline, Week 28 and Week 52
Population: Full Analysis Set - Observed
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 101 | 103
Scores on a Scale
  Week 28 (n=96,103): number analyzed (Participants) | 96 | 103
  Week 28 (n=96,103) | 7.2 (23.94) | 8.4 (26.85)
  Week 52 (n=101,101): number analyzed (Participants) | 101 | 101
  Week 52 (n=101,101) | 7.4 (27.94) | 6.7 (27.84)

42. Secondary Outcome: Change From Baseline at Week 28 and Week 52 in Patient Reported Outcomes (Visual Function Questionnaire-25) - Dependency
Description: as for outcome 35
Time Frame: Baseline, Week 28 and Week 52
Population: Full Analysis Set - Observed
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 101 | 103
Scores on a Scale
  Week 28 (n=96,103): number analyzed (Participants) | 96 | 103
  Week 28 (n=96,103) | 3.3 (27.90) | 9.2 (29.86)
  Week 52 (n=101,101): number analyzed (Participants) | 101 | 101
  Week 52 (n=101,101) | 5.2 (30.77) | 5.7 (33.73)

43. Secondary Outcome: Change From Baseline at Week 28 and Week 52 in Patient Reported Outcomes (Visual Function Questionnaire-25) - Driving
Description: as for outcome 35
Time Frame: Baseline, Week 28 and Week 52
Population: Full Analysis Set - Observed
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 28 | 22
Scores on a Scale
  Week 28 (n=22,22): number analyzed (Participants) | 22 | 22
  Week 28 (n=22,22) | -3.4 (11.69) | 9.8 (23.09)
  Week 52 (n=28,21): number analyzed (Participants) | 28 | 21
  Week 52 (n=28,21) | 0.1 (10.91) | 6.0 (23.59)

44. Secondary Outcome: Change From Baseline at Week 28 and Week 52 in Patient Reported Outcomes (Visual Function Questionnaire-25) - Color Vision
Description: as for outcome 35
Time Frame: Baseline, Week 28 and Week 52
Population: Full Analysis Set - Observed
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 101 | 103
Scores on a Scale
  Week 28 (n=94,100): number analyzed (Participants) | 94 | 100
  Week 28 (n=94,100) | 2.4 (17.22) | 3.0 (19.87)
  Week 52 (n=96,92): number analyzed (Participants) | 96 | 92
  Week 52 (n=96,92) | 4.2 (17.27) | 3.3 (17.47)

45. Secondary Outcome: Change From Baseline at Week 28 and Week 52 in Patient Reported Outcomes (Visual Function Questionnaire-25) - Peripheral Vision
Description: as for outcome 35
Time Frame: Baseline, Week 28 and Week 52
Population: Full Analysis Set - Observed
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 101 | 103
Scores on a Scale
  Week 28 (n=96,103): number analyzed (Participants) | 96 | 103
  Week 28 (n=96,103) | 3.9 (14.20) | 7.5 (20.96)
  Week 52 (n=101,101): number analyzed (Participants) | 101 | 101
  Week 52 (n=101,101) | 3.5 (19.69) | 7.7 (19.92)

46. Secondary Outcome: Change From Baseline at Week 28 and Week 52 in Patient Reported Outcomes (Visual Function Questionnaire-25) - General Health Rating
Description: as for outcome 35
Time Frame: Baseline, Week 28 and Week 52
Population: Full Analysis Set - Observed
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 101 | 103
Scores on a Scale
  Week 28 (n=96,103): number analyzed (Participants) | 96 | 103
  Week 28 (n=96,103) | 3.1 (26.47) | 2.2 (26.91)
  Week 52 (n=101,101): number analyzed (Participants) | 101 | 101
  Week 52 (n=101,101) | 4.2 (26.24) | -0.2 (26.34)

47. Secondary Outcome: Brolucizumab Serum Concentration
Description: To confirm the systemic brolucizumab exposure in a subset of patients.
Time Frame: Approximately 24 hours post Day 1 treatment and approximately 24 hours post Week 24 treatment
Population: Safety Set. Patients in the Safety set with a valid value for the outcome measure.
  Analysis for Weeks 4, 12, 24, 36 and 52 were below the level of quantification (BLQ).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 13 | 0
ng/mL
  Day 2 | 21.1 (4.40) |
  Week 24 + 1 Day (n=7,0): number analyzed (Participants) | 7 | 0
  Week 24 + 1 Day (n=7,0) | 13.4 (4.81) |

48. Secondary Outcome: Number (%) of Patients Who Have Positive Anti-drug Antibody (ADA) Status in Brolucizumab Arm
Description: To assess the immunogenicity of brolucizumab
Time Frame: Up to Week 52
Population: Safety Set. Patients in the Safety set with a valid value for the outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 85 | 0
Participants
  ADA negative (ADA Negative or titer value of 40 at pre-dose) (n=64,0): number analyzed (Participants) | 64 | 0
  ADA negative (ADA Negative or titer value of 40 at pre-dose) (n=64,0) | 35 |
  ADA positive with no boost (ADA Positive at pre-dose) (n=85,0) | 73 |
  Induced (ADA Negative at pre-dose) (n=46,0): number analyzed (Participants) | 46 | 0
  Induced (ADA Negative at pre-dose) (n=46,0) | 16 |
  Boosted (ADA Positive at pre-dose) (n=85,0) | 7 |

49. Secondary Outcome: Ocular Adverse Events (AEs) (>=2% in Any Treatment Arm) by Preferred Term for the Study Eye
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject
Time Frame: Adverse events are reported from first dose of study treatment until end of study treatment plus 30days post treatment, up to a maximum duration of approximately 52 weeks.
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
Participants
  Number of subjects with at least one AE | 57 | 47
  Visual acuity reduced | 12 | 6
  Intraocular pressure increased | 8 | 9
  Meibomian gland dysfunction | 8 | 9
  Cataract | 8 | 3
  Conjunctival haemorrhage | 7 | 5
  Vitreous opacities | 4 | 0
  Dry eye | 3 | 3
  Epiretinal membrane | 3 | 2
  Eye pruritus | 3 | 1
  Uveitis | 3 | 0
  Vitreous haemorrhage | 3 | 5
  Xerophthalmia | 2 | 5

50. Secondary Outcome: Number of Subjects With Non-ocular Adverse Events (AEs) (>=2% in Any Treatment Arm)
Description: as for outcome 49
Time Frame: as for outcome 49
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
Participants | 94 | 74

51. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths are reported from first dose of study treatment until end of study treatment plus 4 weeks post treatment, up to a maximum timeframe of approximately 52 weeks. Post-treatment deaths are reported for the timeframe of greater than 30 days after last treatment, until study completion, up to Week 52. All deaths refer to the sum of on-treatment and post-treatment deaths.
Time Frame: On-treatment - up to 52 weeks; Post-treatment - greater than 30 days after last treatment, until study completion, up to Week 52
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 132 | 131
Participants
  On-Treatment Deaths | 0 | 0
  Post-Treatment Deaths | 0 | 1
  All Deaths | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events are reported from first dose of study treatment until end of study, up to a maximum duration of approximately 52 weeks.
Groups:
- Brolucizumab 6mg: 5 x every 6 weeks loading then every 12 weeks or every 8 weeks maintenance
- Aflibercept 2mg: 5 x every 4 weeks loading then every 8 weeks maintenance
- Overall: Overall
Arm/Group | Brolucizumab 6mg | Aflibercept 2mg | Overall
All-Cause Mortality (participants affected / at risk) | 0/132 | 1/131 | 1/263
Serious Adverse Events (participants affected / at risk) | 28/132 | 22/131 | 50/263
Other Adverse Events (participants affected / at risk) | 92/132 | 84/131 | 176/263
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6mg (N=132) | Aflibercept 2mg (N=131) | Overall (N=263)
Angina unstable (Cardiac disorders) | 0 | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Thyroid mass (Endocrine disorders) | 2 | 0 | 2
Cataract - Fellow eye (Eye disorders) | 5 | 1 | 6
Cataract - Study eye (Eye disorders) | 2 | 2 | 4
Cataract nuclear - Study eye (Eye disorders) | 0 | 1 | 1
Diabetic retinal oedema - Fellow eye (Eye disorders) | 0 | 1 | 1
Retinal artery occlusion - Study eye (Eye disorders) | 1 | 0 | 1
Vitreous haemorrhage - Study eye (Eye disorders) | 0 | 1 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 1
Contrast media allergy (Immune system disorders) | 0 | 1 | 1
Endophthalmitis - Study eye (Infections and infestations) | 1 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Traumatic intracranial haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cerebral infarction (Nervous system disorders) | 2 | 2 | 4
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 2 | 0 | 2
Neuritis (Nervous system disorders) | 1 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 3 | 0 | 3
Diabetic nephropathy (Renal and urinary disorders) | 1 | 3 | 4
End stage renal disease (Renal and urinary disorders) | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Blood pressure inadequately controlled (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1
Subclavian artery stenosis (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6mg (N=132) | Aflibercept 2mg (N=131) | Overall (N=263)
Anaemia (Blood and lymphatic system disorders) | 4 | 4 | 8
Arteriosclerosis coronary artery (Cardiac disorders) | 3 | 6 | 9
Thyroid mass (Endocrine disorders) | 2 | 4 | 6
Cataract - Fellow eye (Eye disorders) | 5 | 0 | 5
Cataract - Study eye (Eye disorders) | 6 | 2 | 8
Conjunctival haemorrhage - Fellow eye (Eye disorders) | 3 | 0 | 3
Conjunctival haemorrhage - Study eye (Eye disorders) | 7 | 5 | 12
Diabetic retinal oedema - Fellow eye (Eye disorders) | 4 | 11 | 15
Diabetic retinopathy - Fellow eye (Eye disorders) | 4 | 1 | 5
Dry eye - Fellow eye (Eye disorders) | 2 | 3 | 5
Dry eye - Study eye (Eye disorders) | 3 | 3 | 6
Epiretinal membrane - Study eye (Eye disorders) | 3 | 2 | 5
Eye pruritus - Fellow eye (Eye disorders) | 3 | 0 | 3
Eye pruritus - Study eye (Eye disorders) | 3 | 1 | 4
Macular oedema - Fellow eye (Eye disorders) | 3 | 1 | 4
Meibomian gland dysfunction - Fellow eye (Eye disorders) | 8 | 9 | 17
Meibomian gland dysfunction - Study eye (Eye disorders) | 8 | 9 | 17
Uveitis - Study eye (Eye disorders) | 3 | 0 | 3
Visual acuity reduced - Fellow eye (Eye disorders) | 10 | 8 | 18
Visual acuity reduced - Study eye (Eye disorders) | 12 | 6 | 18
Vitreous haemorrhage - Study eye (Eye disorders) | 3 | 4 | 7
Vitreous opacities - Fellow eye (Eye disorders) | 4 | 0 | 4
Vitreous opacities - Study eye (Eye disorders) | 4 | 0 | 4
Xerophthalmia - Fellow eye (Eye disorders) | 2 | 8 | 10
Xerophthalmia - Study eye (Eye disorders) | 2 | 5 | 7
Chronic gastritis (Gastrointestinal disorders) | 4 | 1 | 5
Constipation (Gastrointestinal disorders) | 2 | 5 | 7
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 4
Pyrexia (General disorders) | 3 | 2 | 5
Hepatic cyst (Hepatobiliary disorders) | 0 | 3 | 3
COVID-19 (Infections and infestations) | 5 | 1 | 6
Herpes zoster (Infections and infestations) | 4 | 1 | 5
Nasopharyngitis (Infections and infestations) | 3 | 1 | 4
Pneumonia (Infections and infestations) | 0 | 5 | 5
Upper respiratory tract infection (Infections and infestations) | 9 | 9 | 18
Urinary tract infection (Infections and infestations) | 3 | 4 | 7
Alanine aminotransferase increased (Investigations) | 3 | 0 | 3
Bacterial test positive (Investigations) | 3 | 0 | 3
Blood cholesterol increased (Investigations) | 1 | 3 | 4
Blood creatinine increased (Investigations) | 2 | 4 | 6
Blood pressure increased (Investigations) | 6 | 3 | 9
Blood triglycerides increased (Investigations) | 3 | 2 | 5
Blood urea nitrogen/creatinine ratio increased (Investigations) | 3 | 2 | 5
Blood uric acid increased (Investigations) | 4 | 3 | 7
Gamma-glutamyltransferase increased (Investigations) | 3 | 1 | 4
Haemoglobin decreased (Investigations) | 3 | 2 | 5
Intraocular pressure increased - Fellow eye (Investigations) | 3 | 2 | 5
Intraocular pressure increased - Study eye (Investigations) | 8 | 9 | 17
Protein urine present (Investigations) | 6 | 3 | 9
White blood cells urine positive (Investigations) | 4 | 4 | 8
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 7 | 4 | 11
Hyperlipidaemia (Metabolism and nutrition disorders) | 10 | 9 | 19
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 6 | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 0 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 3 | 6
Hypoproteinaemia (Metabolism and nutrition disorders) | 3 | 4 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 4
Carotid arteriosclerosis (Nervous system disorders) | 4 | 4 | 8
Cerebral infarction (Nervous system disorders) | 1 | 3 | 4
Diabetic neuropathy (Nervous system disorders) | 4 | 4 | 8
Headache (Nervous system disorders) | 4 | 1 | 5
Diabetic nephropathy (Renal and urinary disorders) | 4 | 7 | 11
Renal cyst (Renal and urinary disorders) | 4 | 2 | 6
Renal failure (Renal and urinary disorders) | 5 | 1 | 6
Renal impairment (Renal and urinary disorders) | 5 | 1 | 6
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 11
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 | 1 | 4
Eczema (Skin and subcutaneous tissue disorders) | 4 | 1 | 5
Aortic arteriosclerosis (Vascular disorders) | 3 | 1 | 4
Hypertension (Vascular disorders) | 7 | 12 | 19
Peripheral arterial occlusive disease (Vascular disorders) | 3 | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/67/NCT04058067/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT04058067/SAP_001.pdf